CLINICAL TRIAL: NCT01864200
Title: A Randomized, Double-Blind, Placebo-Controlled Study Comparing CroFab® vs Placebo With Rescue Treatment for Copperhead Snake Envenomation
Brief Title: Randomized, Double-Blind, Placebo-Controlled Study: CroFab® vs Placebo for Copperhead Snake Envenomation
Acronym: Copperhead
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: BTG International Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BTG-PR005-002
Record Dates: First submitted 2013-05-24; First posted 2013-05-29 (Estimated); Results first posted 2017-11-22 (Actual); Last update posted 2017-11-22 (Actual); Status verified 2017-10

CONDITIONS: Snake Bites
MeSH Terms: conditions — Snake Bites | interventions — Crotalidae Polyvalent immune Fab; Red Meat

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CroFab (Experimental): crotalidae polyvalent immune fab (ovine) per approved labeling
  Interventions: Biological: Crotalidae polyvalent immune fab (ovine)
- Saline placebo (Placebo Comparator): Saline placebo
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Crotalidae polyvalent immune fab (ovine) — crotalidae antivenom
  Other Names: CroFab
  Arms: CroFab
Biological: Placebo — Saline placebo
  Arms: Saline placebo

SUMMARY:
This study will evaluate the recovery from copperhead snake bite in patients with mild or moderate venom effect. Potential subjects received CroFab antivenom or placebo. After blinded treatment and discharge, the subject returns to the clinic for follow-up assessments at day 3, 7, 14, and 28 after snake bite as well as follow-up telephone assessments on day 10, 17, and 24 after snake bite. The purpose of this study is to compare recovery in copperhead snake bite patients treated with antivenom vs placebo (no active drug) as measured by the Patient Specific Functional Scale (PSFS) at Day 14 follow-up. The primary efficacy endpoint of this study was achieved.

DETAILED DESCRIPTION:
This study will evaluate the recovery from copperhead snake bite in patients with mild or moderate venom effect. Potential subjects will receive CroFab antivenom or placebo. The trial is conducted by emergency room doctors, toxicologists, or surgeons at hospitals in regions where copperhead bites are common. After blinded treatment and discharge, the subject returns to the clinic for follow-up assessments at day 3, 7, 14, and 28 after snake bite. The subject will also be called by telephone for follow-up assessments on day 10, 17, and 24 after snake bite. The purpose of this study is to compare recovery in copperhead snake bite patients treated with antivenom vs placebo (no active drug) as measured by the Patient Specific Functional Scale (PSFS) at Day 14 follow-up.The primary efficacy endpoint of this study was achieved. Treatment with CroFab® demonstrated measurable and significant improvement (less disability) over placebo: in the mITT population, the LS mean total score on the PSFS at Day 14 follow-up and treatment showed less disability in patients randomized to receive CroFab® than those receiving placebo.

ELIGIBILITY:
Inclusion Criteria-

* Envenomation by a copperhead snake

  a. Snake identified by one of the following means: i.Snake or photograph of snake brought to Emergency Department ii.Patient chooses copperhead from an array of snake photographs iii.Patient envenomated in an area where only copperheads are endemic iv.Patient envenomated by a captive copperhead snake
* Completion of informed consent and eligibility confirmation within 24 hours of envenomation
* Envenomation on only one extremity, distal to the elbow or knee
* Clinical evidence of mild or moderate venom effect (limb swelling and/or tenderness) is present (Venom effects need not be progressing.)
* Patient willing and able to complete follow-up schedule of assessments
* Patient is able to read, comprehend and sign the IRB approved consent document(s)
* Patient is able to read and comprehend the written assessment tools (e.g., DASH, LEFS, PROMIS Physical Function Short Form 10a (PROMIS PF-10), PGIC, etc.)
* Patient is ≥12 years of age
* Patient is sober, competent, and able to complete verbal and written informed consent

Exclusion Criteria-

* Patient has clinical evidence of severe venom effect as defined by meeting any one of the following parameters:

  i. Swelling to an entire extremity (all major joints affected)
  1. Lower extremity: swelling crossing hip joint
  2. Upper extremity: swelling crossing shoulder joint ii. INR > 2.0 iii. Platelets <50,000 cells / µL iv. Fibrinogen <50 mg/dL

  v. Compartment syndrome vi. Systolic Blood Pressure <90 mmHg vii. More than minimal bleeding viii. Investigator's clinical discretion
* Patient has already received antivenom for the management of the current envenomation
* Patient is pregnant or breastfeeding
* Patient is a prisoner
* Patient has a distracting injury or condition with acute pain or functional impairment, and/or is unable to make a reliable self-report of functionality status based solely on the condition of interest
* Patient had a previous snake envenomation to any body area in the 30 days prior to screening/enrollment, regardless of whether antivenom was administered for the previous envenomation
* Patient had an acute traumatic event, surgery, an acute medical event, or exacerbation of a pre-existing medical or surgical condition affecting the envenomated extremity within the 30 days prior to screening/enrollment
* Patient has participated in a clinical study involving an investigational pharmaceutical product or device within the 3 months prior to screening that may have impact on clinical outcomes of snakebite
* Patient has previously participated in this clinical study
* Patient has a known history of hypersensitivity to any components of CroFab®, or to papaya or papain
* Patient is otherwise unsuitable for inclusion in this study, based on the opinion of the Investigator

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2013-07; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maria Gasior, MD, Principal Investigator — BTG International Inc.
Locations (18):
- United States (18):
  - Georgia Regents University, Augusta, Georgia
  - University of Kansas Hospital, Kansas City, Kansas
  - Washington University, St Louis, Missouri
  - University of North Carolina, Chapel Hill, North Carolina
  - Duke University, Durham, North Carolina
  - Vidant Medical Center, Greenville, North Carolina
  - Lehigh Valley Hospital Center, Allentown, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Palmetto Health Richland, Columbia, South Carolina
  - St Joseph Regional Health Center, Bryan, Texas
  - University of Texas - Southwestern, Dallas, Texas
  - Ben Taub General Hospital, Houston, Texas
  - Texas Children's Hospital, Houston, Texas
  - Scott & White Hospital, Temple, Texas
  - University of Virginia, Charlottesville, Virginia
  - Virginia Commonwealth University, Richmond, Virginia
  - Marshall Health, Huntington, West Virginia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- CroFab: crotilidae polyvalent immune fab (ovine) per approved labeling
  crotilidae polyvalent immune fab (ovine): crotilidae antivenom
- Saline Placebo: Saline placebo
  Placebo
Period: Overall Study
Arm/Group | CroFab | Saline Placebo
Started | 45 | 29
Completed | 43 | 26
Not Completed | 2 | 3
Not completed — Lost to Follow-up | 1 | 3
Not completed — Protocol Violation | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CroFab | Saline Placebo | Total
Number analyzed (Participants) | 45 | 29 | 74
Age, Continuous [Mean (Standard Deviation); unit: years] | 44 (17.9) | 42 (17.2) | 43.04 (17.57)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 13 | 35
  Male | 23 | 16 | 39
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 2 | 4
  White | 40 | 25 | 65
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 2 | 4
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 45 | 29 | 74

OUTCOME MEASURES:

1. Primary Outcome: Patient Specific Functional Scale Score
Description: Patient Specific Functional Scale (PSFS) at 14 day follow-up This is a three-item instrument, administered verbally, that is used to evaluate whether a health condition impacts a patient's ability to perform activities that are important to him/her. On the initial assessment, the patient is asked to identify "up to three important activities that you are unable to do or are having difficulty with as a result of your (snakebite)." The patient then provides a rating for each item, on an 11-point ordinal scale ranging from 0 ("unable to perform activity") to 10 ("able to perform activity at the same level as before the injury or problem"). During reassessments, the subject is prompted to re-rate the same three activities. The average of up to 3 specific activity scores was recorded, and the range of possible scores is 0 - 10. Higher scores indicate less impairment.
Time Frame: at 14 day follow-up
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | CroFab | Saline Placebo
Number analyzed (Participants) | 45 | 28
units on a scale | 8.62 (0.550) | 7.45 (0.603)

ADVERSE EVENTS:
Time Frame: Envenomation + 28 days
Arm/Group | CroFab | Saline Placebo
Serious Adverse Events (participants affected / at risk) | 1/45 | 1/29
Other Adverse Events (participants affected / at risk) | 25/45 | 8/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CroFab (N=45) | Saline Placebo (N=29)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Venom poisoning (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CroFab (N=45) | Saline Placebo (N=29)
Dizziness (Nervous system disorders) | 4 (4) | 2 (3)
Headache (Nervous system disorders) | 5 (8) | 1 (1)
Paraesthesia (Nervous system disorders) | 3 (3) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 5 (5) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 5 (5) | 0 (0)
Pyrexia (General disorders) | 4 (4) | 0 (0)
Nausea (Gastrointestinal disorders) | 4 (4) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (4) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No